CLINICAL TRIAL: NCT01547910
Title: Effect of Supplementation of Fish Oil on Non-alcoholic Fatty Liver Disease in Children - a Randomized, Double Blind, Placebo Controlled, Multicenter Study
Brief Title: Effect of Supplementation of Fish Oil on Non-alcoholic Fatty Liver Disease in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Piotr Socha (Other)
Collaborators: Medical University of Bialystok (Other); Medical University of Silesia (Other); Pediatric Municipal Hospital of Rzeszow, Poland (Unknown)
Responsible Party: Sponsor-Investigator, Piotr Socha, Professor PhD MD, Principal Investigator, Children's Memorial Health Institute, Poland
Organization: Children's Memorial Health Institute, Poland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ChildrensMHIPoland
Record Dates: First submitted 2012-02-29; First posted 2012-03-08 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: fatty liver; hepatitis; insulin resistance; unsaturated fatty acids; NAFLD, children
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Hepatitis; Insulin Resistance | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish oil (Experimental): Children will receive fish oil capsules according to age as described in the protocol
  Interventions: Dietary Supplement: Fish Oil
- Placebo (Placebo Comparator): Sunflower oil in the same capsules (the same shape and colour) given in the same regime as 'fish oil' capsules
  Interventions: Dietary Supplement: Fish Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — Fish oil given in supplementary dose

SUMMARY:
The aim of this study is to evaluate efficacy of fish oil (EPA/DHA) in children with non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
76 children or adolescents aged 6-19 with NAFLD will be included in the study. Diagnosis of NAFLD is set by increased alanine transaminase and features of liver steatosis on ultrasound. Patients will be randomized to receive either fish oil (EPA/DHA, 400-1200mg) or placebo (sunflower oil) for 6 months. All children will be advised to reduce weight (dietetic intervention + increased physical activity). Laboratory tests, liver ultrasound, anthropometric analysis will be performed at the start, after 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* age 6-19
* overweight or obesity
* ALT activity over 130% of upper limit norm
* hyperechogenicity of the liver on ultrasound

Exclusion Criteria:

* HCV, HBV infection
* cholestasis
* chronic/acute liver failure
* alpha-1-antitrypsin deficiency
* Wilson disease
* type 2 diabetes mellitus
* beta-oxidation defects
* alcohol consumption
* history of parenteral nutrition
* use of drugs

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2007-08; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Serum alanine transaminase level decrease min. 0.3 upper limit of normal | 6 months
  Number of patients in whom ALT decreased min. 0.,3 ULN in 'fish oil' group compared to 'placebo' group

SECONDARY OUTCOMES:
normalization of liver imaging on ultrasound | after 6 months of therapy
  'Fish oil' group will be compared to 'placebo' group
ALT and AST activity | 6 months
  'Fish oil' group will be compared to 'placebo' group
Insulin resistance markers as Homa-IR | 6 months
  'Fish oil' group will be compared to 'placebo' group
Fat and lean body mass measurements | 6 months
  'Fish oil' group will be compared to 'placebo' group
Caloric intake including fat intake and sucrose intake | 6 months
  'Fish oil' group will be compared to 'placebo' group

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Socha, Principal Investigator — Children's Memorial Health Institute, Warsaw, Poland

REFERENCES:
- [Derived] Janczyk W, Lebensztejn D, Wierzbicka-Rucinska A, Mazur A, Neuhoff-Murawska J, Matusik P, Socha P. Omega-3 Fatty acids therapy in children with nonalcoholic Fatty liver disease: a randomized controlled trial. J Pediatr. 2015 Jun;166(6):1358-63.e1-3. doi: 10.1016/j.jpeds.2015.01.056. Epub 2015 Mar 11. PMID 25771388
- [Derived] Janczyk W, Socha P, Lebensztejn D, Wierzbicka A, Mazur A, Neuhoff-Murawska J, Matusik P. Omega-3 fatty acids for treatment of non-alcoholic fatty liver disease: design and rationale of randomized controlled trial. BMC Pediatr. 2013 May 23;13:85. doi: 10.1186/1471-2431-13-85. PMID 23702094